CLINICAL TRIAL: NCT05746117
Title: Continual vs. Routine Home Blood Pressure Monitoring and Management in Diverse Community Practice: CHANGE-BP
Acronym: CHANGE-BP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study aborted by the sponsor
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBPM_CHANGE-BP2022
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
Keywords: Hypertension; Medical Device
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Continuous Blood Pressure Monitoring (CBPM) (Experimental): Participants will wear the Aktiia Bracelet for 6-months and potentially receive blood pressure medication titrations during the 6-month period.
  Interventions: Device: Aktiia Device
- Home Blood Pressure Monitoring (HBPM) (Active Comparator): Participants will receive an upper arm cuff and standard hypertension care from their primary care physician.
  Interventions: Device: Upper arm cuff

INTERVENTIONS:
Device: Aktiia Device — The Aktiia Bracelet is a CE-marked medical device that will be used in accordance with its instructions for use. The bracelet non-invasively measures optical signals at the wrist, which are used to determine blood pressure. The bracelet comes with a bluetooth enabled upper arm cuff that can be used to take on-demand blood pressure measurements. All measurements are transmitted to a dashboard that a clinical pharmacist monitors during the participant's enrollment in the study.
  Arms: Continuous Blood Pressure Monitoring (CBPM)
Device: Upper arm cuff — A standard upper arm oscillometric cuff that can be used to take blood pressure at home.
  Arms: Home Blood Pressure Monitoring (HBPM)

SUMMARY:
The purpose of the CHANGE-BP study is to examine the change in in-office measured Blood Pressure (BP) from baseline to end of study (6-months) between participants randomized to either 1) Continual Blood Pressure Monitoring (CBPM), which includes receiving Aktiia's novel cuffless BP Research System that has an accompanying Aktiia Patient Interface smartphone application, and care delivered through a centralized Aktiia Provider Interface that displays device data and is accessible by a health care professional or 2) Home Blood Pressure Monitoring (HBPM), which includes a standard oscillometric blood pressure cuff and the standard blood pressure management care from a participant's primary care physician.

DETAILED DESCRIPTION:
This is a prospective, unblinded, open-label, randomized clinical trial that will study the use of the investigational Aktiia Bracelet and an accompanying Provider Interface in hypertension management. The Aktiia Bracelet is a non-invasive blood pressure monitor intended to track systolic and diastolic blood pressure and heart rate.

Participants will attend a baseline visit, which will include a survey and blood pressure and anthropometric measurements. Participants will then be randomized to either the CBPM group, which includes the Aktiia Bracelet and care through a centralized Aktiia Provider Interface, or the HBPM group, which includes a standard blood pressure cuff and standard hypertension care. Individuals in the CBPM group will wear the Aktiia Bracelet for 6 months. During this time, a study-affiliated clinical pharmacist will monitor the individual's blood pressure through the Provider Interface and will potentially titrate the participant's blood pressure medications accordingly. After 6-months, all participants will return for an end of study visit that will include a survey and blood pressure and anthropometric measurements. Participants in the CBPM group will complete an additional survey to give their opinion on the Aktiia product.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 years old
* Owns a smartphone that is an Android or iOS with a data plan
* Fluent in written and spoken English as the technology is currently only available in English
* Average of 3 BP readings in last 18 months of >140/90 OR last in-office BP >140/90 in the last 6 months as documented in their Electronic Health Record
* Is a patient with Providence Health
* Willing to attend the 2 in-person study visits
* Is not participating in another study that is designed to influence blood pressure
* Willing to wear the Aktiia bracelet for 6 months
* Willing to be randomized to either group
* Had a BMP in the last 12 months or is willing to get one at the discretion of the clinical pharmacist as standard of care

Exclusion Criteria:

* Blood pressure at the baseline in-office visit is too low (SBP <140 mmHg AND DBP <90 mmHg) OR is too high (SBP > 190 mmHg OR DBP > 120 mmHg)
* Tachycardia (heart rate at rest > 120bpm)
* Atrial fibrillation, persistent or chronic
* Cardiomyopathy with LVEF <40% documented within the past year
* Diabetes Mellitus
* Under active treatment for hyperthyroidism
* Myxedema coma
* Subclavian stenosis
* Pheochromocytoma
* Raynaud's disease
* Trembling and shivering
* Known pregnancy
* Breastfeeding
* Arteriovenous fistula
* Arm amputation
* Exfoliative skin disease
* Lymphedema
* Known allergy to silicone
* Terminal medical condition with a life expectancy less than 2 years
* CKD 4-5 (eGFR ≤ 30 mL/min)
* Upper arm circumference < 22 cm or > 42 cm
* Wrist circumference < 14 cm or > 21 cm
* Adults unable to consent or who need a legally authorized representative to consent
* Currently incarcerated or detained in accordance with federal regulations regarding prisoners (e.g., 45 CFR 46 Subpart C)
* Diagnosed whitecoat hypertension
* On hospice or going on hospice in the next 6-months
* Currently undergoing or will undergo active IV infusions for chemotherapy
* Any condition which, at the discretion of the enrolling investigator, would preclude their ability to comply with study procedures

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | 6-months
  Determine if there is a statistically greater reduction in in-office measured blood pressure from baseline to 6-months in the CBPM arm when compared to the HBPM arm

SECONDARY OUTCOMES:
Participant perception | 6-months
  Statistics on participants' perception of an optical BP monitoring modality as compared to an oscillometric cuff
Participant engagement | 6-months
  Statistics on participants' engagement with the Aktiia Research System over the 6-month period
Participant compliance | 6-months
  Statistics on participants' compliance, which is operationalized as the number of measurements made each day by the Aktiia Research System and the number of times the user syncs their Aktiia bracelet with the Patient Interface for the CBPM arm. Statistics on the number of upper arm cuff measurements reported to their PCP in the HBPM arm.
Participant sociodemographics | 6-months
  Statistics on the sociodemographic breakdown of the sample

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Shoenkerman, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Health & Services, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No